CLINICAL TRIAL: NCT01894893
Title: Atlas of Human Milk Nutrients
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 11.33.NRC
Record Dates: First submitted 2013-04-25; First posted 2013-07-10 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Breastfeeding Mothers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Mother milk
  2. Umbilical cord blood
  3. Mother blood
  4. Adipose tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breastfeeding mothers

SUMMARY:
The main objective of this clinical trial is to collect human milk samples from 0 to 4 months after delivery in order to characterize human milk components. The secondary objectives of this study are:

1. To assess whether there is a correlation between human milk composition and mothers' diet
2. To assess whether there is a correlation between human milk composition and maternal clinical parameters
3. To assess whether there is a correlation between human milk composition and mother and infant clinical parameters

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years of age included at time of enrolment
* BMI before pregnancy between 19 and 29 included
* Having signed the Informed Consent Form
* Having decided to exclusively breast-feed until infant is 4 months old

Exclusion Criteria:

* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study
* Presenting any disease or medical condition which might prevent breast-feeding or collection the human milk samples or for which breast-feeding is not indicated
* Presenting diseases/medical conditions such as diabetes, heart problems, abnormal conditions of pregnancy (ex. hypertension)
* Presenting dietary problems/illnesses such as anorexia, bulimia and celiac disease
* Assuming any medication indicated for the treatment of any metabolic or cardiovascular disease
* Cannot be expected to comply with the study procedures

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy mothers of any ethnicity having decided to exclusively breast-feed their new born baby from birth up to 4 months of age will be eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Characterization of human milk components | Between 0 and 4 months after delivery
  Nutrients in human breast milk samples will be characterized and quantified by analysing with modern analytical techniques (NMR, HPLC-MS and GC-MS) the human milk samples collected at each study visits (3d, 14 days, 1m, 2m, 3m and 4 months after delivery, 1 week after delivery, ). The parameters which will be assessed in human milk samples are : Total Energy Value, Total Macronutrients (lipids, proteins, carbohydrates, solids), Lipids' characterization, Peptide profiling, Oligosaccharides profiling, and Micro-RNA profiling. It will be done in 240 completed mothers.

SECONDARY OUTCOMES:
Human milk composition versus mothers' diet data | between 3 months before delivery and 4 months after delivery
  The human milk composition profiles (primary outcome) will be correlated in a longitudinal manner to mothers' diet. Information on mother's diet will be collected using a 3-days diary and entering the data in Nutrilog (total intake of the mothers). This will be done before each study visit in 240 completed mothers.
Human milk composition versus maternal clinical parameters | Between 0 and 4 months after delivery
  The human milk composition profiles will be correlated in a longitudinal manner to the stage of lactation, the gestation's age, the type of delivery, the sex of the baby, the number of babies the mother already had (gravidity and parity), single/multiple birth. It will be done in 240 completed mothers.
Human milk composition versus mother and infant clinical parameters | Between 0 and 4 months after delivery
  The human milk composition profiles will be correlated in a longitudinal manner to infant anthropometric measurements (weight, height and head circumference). It will be done in 240 completed mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Billeaud, Prof, Principal Investigator — University Hospital, Bordeaux; Jean-Charles Picaud, Prof, Principal Investigator — Hôpital de la Croix-Rousse; Thameur Rakza, Dr, Principal Investigator — CHRU de Lille; Massimo Agosti, Dr, Principal Investigator — Ospedale del Ponte Varese; Tom Stiris, Dr, Principal Investigator — Oslo University Hospital; Silva Gorett, Dr, Principal Investigator — Hospital de S. João Porto; Almerinda Barroso Pereira, Dr, Principal Investigator — Hospital de São Marcos - Braga; Maria Jose Costeira, Dr, Principal Investigator — Guimarães Hospital Braga; Isam Al-Jashi, Dr, Principal Investigator — Al Jashi Isam Private Med. Practice Bucharest; Sylvia Stoicescu, Dr, Principal Investigator — Polizu Hospital Bucharest; Cecilia Martinez-Costa, Dr, Principal Investigator — Hospital Clínico Universitario de Valencia; Magnus Domellöf,, Dr, Principal Investigator — Umeå University; Mireille Vanpeé, Dr, Principal Investigator — Karolinska University hospital in Solna; Giovanna Marchini, Dr, Principal Investigator — Karolinska University hospital in Solna
Locations (13):
- France (3):
  - CHU Bordeaux, Bordeaux
  - CHRU de Lille, Lille
  - Hôpital de la Croix Rousse, Lyon
- Ospedale del Ponte, Varese, Italy
- Oslo University Hospital, Oslo, Norway
- Portugal (3):
  - Centro Hospitalar do Alto Ave Guimarães Hospital, Braga
  - Hospital de São Marcos, Braga
  - Hospital de S. João, Porto
- Romania (2):
  - Al Jashi Isam Private Med. Practice, Bucharest
  - Polizu Hospital, Bucharest
- Hospital Clínico Universitario de Valencia, Valencia, Spain
- Sweden (2):
  - Department of Woman and Child Health, Karolinska University Hospital, Stockholm, Stockholm County
  - Umeå University hospital, Umeå

REFERENCES:
- [Derived] Raymond F, Lefebvre G, Texari L, Pruvost S, Metairon S, Cottenet G, Zollinger A, Mateescu B, Billeaud C, Picaud JC, Silva-Zolezzi I, Descombes P, Bosco N. Longitudinal Human Milk miRNA Composition over the First 3 mo of Lactation in a Cohort of Healthy Mothers Delivering Term Infants. J Nutr. 2022 Jan 11;152(1):94-106. doi: 10.1093/jn/nxab282. PMID 34510208
- [Derived] Binia A, Lavalle L, Chen C, Austin S, Agosti M, Al-Jashi I, Pereira AB, Costeira MJ, Silva MG, Marchini G, Martinez-Costa C, Stiris T, Stoicescu SM, Vanpee M, Rakza T, Billeaud C, Picaud JC, Domellof M, Adams R, Castaneda-Gutierrez E, Sprenger N. Human milk oligosaccharides, infant growth, and adiposity over the first 4 months of lactation. Pediatr Res. 2021 Sep;90(3):684-693. doi: 10.1038/s41390-020-01328-y. Epub 2021 Jan 14. PMID 33446921